CLINICAL TRIAL: NCT01907425
Title: Prenatal Molecular Characterisation by CGH+SNP-ARRAY of Supernumerary Marker Chromosomes and de Novo Apparently Balanced Reciprocal Translocations
Acronym: compass
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: futility
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Callier PHRC N 2012
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Pre-natal Patient
MeSH Terms: interventions — Blood Specimen Collection

ARMS (1):
- Pre-natal Patient (Other)
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples

SUMMARY:
In the prenatal period, les supernumerary marker chromosomes (SMC) and de novo apparently balanced reciprocal translocations are revealed by foetal karyotyping, which does not always make it possible to determine whether the anomaly is balanced or not and does not reveal uniparental disomy. The presence of these chromosomal rearrangements raises a difficult question for genetic counselling during pregnancy because of the risk of intellectual deficiency in the foetus. CGH+SNP-Array can provide information concerning 1) the balanced or not nature of these translocations 2) the presence or not of euchromatin in the SMC 3) the presence or not of uniparental disomy.

ELIGIBILITY:
Inclusion Criteria:

* Metaphase karyotyping with SMC or a de novo Apparently-balanced reciprocal translocation
* Parents covered by the National Health Insurance Agency,
* Consent of the parents

Exclusion Criteria:

* Persons not covered by the National Health Insurance Agency
* Normal foetal karyotyping or showing chromosomal anomalies not related to the present study (trisomy 18….) or inherited anomalies
* Absence of a sample from one of the parents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-08-30 (Actual); Primary Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
supernumerary chromosome markers | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France